CLINICAL TRIAL: NCT00069862
Title: Iron Balance Study of DFO and GT56-252 in Patients With Transfusional Iron Overload Secondary to Beta-Thalassemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GTC-134-102
Record Dates: First submitted 2003-10-02; First posted 2003-10-03 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: Beta-Thalassemia
Keywords: Beta Thalassemia
MeSH Terms: conditions — beta-Thalassemia | interventions — 4'-hydroxydesazadesferrithiocin

INTERVENTIONS:
Drug: Deferitrin (GT56-252)
Drug: desferoxamine (DFO)

SUMMARY:
A clinical trial designed to compare the safety and iron excretion properties of desferoxamine (DFO) and deferitrin (GT56-252), an experimental oral iron chelator.

ELIGIBILITY:
Inclusion Criteria:

* Beta-thalassemia patients, 18 years of age or older, currently undergoing chronic blood transfusion therapy and iron chelation therapy who weigh more than 40 kg.
* No clinically significant findings on physical exam, medical history, or screening laboratories.
* Serum ferritin greater than 500 ng/mL, serum creatine creatinine within the normal range and platelet count greater than 100,000/mm3.
* Willing and able to discontinue DFO or L1 for the period of study.
* Woman of child-bearing potential must have a negative serum pregnancy test at screening and use a medically acceptable form of birth control during the study and for 1 month afterward. Male patients must also use barrier contraceptives during the study and for 1 month afterward.
* Have a level of understanding and willingness to cooperate with the confinement and all procedures. Able to provide voluntary signed/dated written informed consent.

Exclusion Criteria:

* Serious medical condition unrelated to Beta-Thalassemia.
* Participation in a previous investigational drug study within 30 days preceding screening.
* Patients with a known allergy to DFO that prevents chronic administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25
Dates: Start 2003-09; Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
safety and tolerability
iron excretion in urine and stool
pharmacokinetic measurements

CONTACTS AND LOCATIONS:
Locations (1):
- The New York Presbyterian Hospital-Weill Medical College of Cornell University, New York, New York, United States